CLINICAL TRIAL: NCT06165991
Title: The Effect of Bupivacaine Liposome Combined With Bupivacaine Hydrochloride on Thoracic Paravertebral Nerve Block for Postoperative Pain After Thoracoscopic Lung Surgery
Brief Title: Liposomal and Standard Bupivacaine in Thoracic Paravertebral Block for Post-Thoracoscopic Pain
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongtao Sun (Other)
Responsible Party: Sponsor-Investigator, Yongtao Sun, Professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: liposomal bupivacaine LB
Record Dates: First submitted 2023-11-29; First posted 2023-12-12 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Thoracic Paravertebral Block; Postoperative Analgesia; Thoracoscopic Lobectomy
Keywords: liposomal bupivacaine(LB); Thoracic paravertebral nerve block; Postoperative analgesia; thoracoscopic lobectomy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: bupivacaine hydrochloride (Active Comparator): Group A: Patients in the control group received 20 mL of 0.5% bupivacaine hydrochloride (total dose, 100 mg).
  Interventions: Drug: Group A: bupivacaine hydrochloride;
- Group B: liposomal bupivacaine and bupivacaine hydrochloride (Experimental): Patients in the intervention group received a mixture of 10 mL of 1.33% liposomal bupivacaine (133 mg) and 10 mL of 0.5% bupivacaine hydrochloride.
  Interventions: Drug: GroupB:Liposomal bupivacaine and bupivacaine hydrochloride;

INTERVENTIONS:
Drug: GroupB:Liposomal bupivacaine and bupivacaine hydrochloride; — Group B::Patients in the intervention group received a mixture of 10 mL of 1.33% liposomal bupivacaine (133 mg) and 10 mL of 0.5% bupivacaine hydrochloride.
  Arms: Group B: liposomal bupivacaine and bupivacaine hydrochloride
Drug: Group A: bupivacaine hydrochloride; — Group A:Patients in the control group received 20 mL of 0.5% bupivacaine hydrochloride (total dose, 100 mg).
  Arms: Group A: bupivacaine hydrochloride

SUMMARY:
I. Research purpose

1.1 Main Objective: To investigate the efficacy and safety of bupivacaine liposome thoracic paravertebral nerve block for postoperative analgesia after thoracoscopic lobectomy

1.2 Exploratory Objective: To investigate the noninferiority of bupivacaine liposomes in thoracic paravertebral nerve block with standard bupivacaine

DETAILED DESCRIPTION:
Standard monitoring, including electrocardiography (ECG), heart rate (HR), noninvasive blood pressure (NIBP), pulse oxygen saturation (SpO2), end-tidal carbon dioxide (ETCo2), and bispectral index (BIS) was initiated on arrival in the operating room. A neuromuscular monitor (JS-100, Beijing SLGO Medical Technology Co., Ltd., China) was used to confirm neuromuscular block (NMB).

Intravenous anesthesia was induced with 0.04 mg/kg midazolam, 0.3-0.5 μg/kg sufentanil, 1.5-2.5 mg/kg propofol, and 0.6 mg/kg rocuronium. Hemodynamics were supported with vasoactive agents (atropine, norepinephrine, dopamine, esmolol) as needed. After the train of four count (TOFC) ratio reached zero, a double-lumen tube or a single-lumen tube with a bronchial blocker was inserted, with correct positioning confirmed by fiberoptic bronchoscopy. Under real-time ultrasound visualization, a senior anesthesiologist performed thoracic paravertebral blocks at the T4-5, T6-7, and T8-9 levels in patients placed in the lateral decubitus position, injecting 6 mL, 8 mL, and 6 mL of local anesthetic at the respective levels.

Group B : Patients in the intervention group received a mixture of 10 mL of 1.33% liposomal bupivacaine (133 mg) and 10 mL of 0.5% bupivacaine hydrochloride,.

Group A: whereas those in the control group received 20 mL of 0.5% bupivacaine hydrochloride (total dose, 100 mg).

All patients received total intravenous anesthesia during surgery. Propofol was administered at a rate of 2-4 mg/kg/h, and remifentanil was administered at a rate of 0.05-0.3 μg/kg/min to maintain a BIS value range from 40 to 60. Rocuronium will be administered and adjusted to achieve deep NMB (defined as a TOFC=0 and a post-tetanic count =1-2). Standard ventilation parameters included a respiratory rate of 10-12 breaths·min-¹ and a positive end-expiratory pressure (PEEP) of 5cmH₂O. During double-lung ventilation, a tidal volume of 8 mL/kg was used, with ETCo2 maintained between 35-45 mmHg and peak airway pressure kept below 20cmH₂O. During single-lung ventilation, the tidal volume was reduced to 6 mL/kg, with ETCo2 maintained below 60 mmHg and peak airway pressure kept below 30cmH₂O. Intravenous sufentanil (0.15 μg/kg) and ondansetron hydrochloride (8mg) were administered prior to the end of surgery. After surgery, patients were transferred to the post-anesthesia care unit (PACU) for further monitoring. Additionally, 2-4 mg/kg of sugammadex was given to reverse the residual effect of rocuronium.

In the PACU, an intravenous bolus of 0.1 μg/kg sufentanil was administered when the numeric rating scale (NRS; 0, no pain; 1-3, mild pain; 4-6, moderate pain; and 7-10, severe pain) score was ≥4. The drugs used for postoperative patient-controlled intravenous analgesia (PCIA) were sufentanil (2 μg/kg), which were diluted in 0.9% normal saline to a final volume of 100mL. The analgesia pump settings were as follows: background dose, 0 mL/h; self-controlled additional dose, 1 mL/time; and lockout time, 10 min. The patients were sent to the ward upon meeting the following criteria for at least 30 minutes: NRS score <4, an Adrelete score ≥9 and absence of other adverse reactions. The number of PCA attempts and the total drug delivery were automatically recorded by the postoperative analgesia system.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old;

  2) Patients undergoing unilateral initial thoracoscopic lobectomy under general anesthesia (TV or robot-assisted);

  3) American Society of Anesthesiologists (ASA) Grade I - III;

  4) Voluntarily participate in the study and sign the informed consent.

Exclusion Criteria:

* 1) Pregnant or lactating women;

  2) Pulmonary wedge-shaped resection;

  3) ≥2 thoracic drainage tubes;

  4) Abnormal liver function: ALT and/or AST>2×ULN, or

TBIL≥1.5×ULN;

5) Renal function impairment (serum creatinine >176μmol/L), or received dialysis treatment within 28 days before surgery;

6) Participate in another research trial involving an investigational drug within 6 months;

7) A history of drug or alcohol abuse;

8) Long-term use of opioids (more than 3 months or more than 5 mg daily morphine equivalent per day for 1 month);

9) History of allergy to local anesthetics or one of the investigational drugs;

10) Uncontrolled mental or neurological symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
area under the NRS score curve (AUC) for resting | 48hours postoperative
  area under the NRS score curve (AUC) for resting and active 48 hours after surgery

SECONDARY OUTCOMES:
15 quality of recovery assessments (QoR15) | at 24, 48, and 72 hours after surgery
  15 quality of recovery assessments (QoR15) at 24, 48, and 72 hours after surgery. Its scores range from 0 to 150, with higher scores indicating better recovery.Based on the scores, QoR can be classified into excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121), and poor (QoR-15 <90).
area under the NRS score curve (AUC) for exercise | 48 hours after surgery
  area under the NRS score curve (AUC) for resting and exercise 48 hours after surgery
area under the NRS score curve (AUC) for resting and exercise | 72 hours after surgery
  area under the NRS score curve (AUC) for exercise 72 hours after surgery
area under the NRS score curve (AUC) for resting and exercise | 96 hours after surgery
  area under the NRS score curve (AUC) for resting and exercise 96 hours after surgery
cumulative opioid consumption (morphine milligram equivalent, MME | at 72 hours after surgery
  cumulative opioid consumption at 72 hours after surgery (morphine milligram equivalent, MME

CONTACTS AND LOCATIONS:
Overall Officials: Sun Y tao, PH.D, Study Chair — Shandong First Medical University
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Sun Y, Guo N, Fang T, Feng Y, Liu P, Sun D, Li Y, Liu K, Ren Y, Li M, Liu Q, Yang X, Chi Y, Liu Z, Yuan L, Lang B, Yang Z, Feng N, You P, Zhang W, Su D, Wu J. Effect of preoperative thoracic paravertebral block using liposomal bupivacaine combined with drainage-tube patient-controlled analgesia on postoperative pain after thoracoscopic lobectomy: a prospective, multicentre, double-blind, randomized controlled study protocol. Perioper Med (Lond). 2025 Nov 6;14(1):122. doi: 10.1186/s13741-025-00564-2. PMID 41199334